CLINICAL TRIAL: NCT03255460
Title: Investigation of the Relationship Between Fatigue and Physical Activity Level in Patients With Multiple Sclerosis
Brief Title: The Relationship Between Fatigue and Physical Activity Level in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, Research Asisstant, Gazi University
Other Study IDs: Gazi 1
Record Dates: First submitted 2017-08-12; First posted 2017-08-21 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Fatigue; Physical Activity; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple Sclerosis individuals: Multiple sclerosis patients included in this study. Inclusion and exclusion criteria were considered.
- Healthy individuals: Those without chronic disease were included in the study. Inclusion and exclusion criteria were considered.

SUMMARY:
Multiple sclerosis (MS) is a chronic, progressive and unpredictable disease of the central nervous system. In MS, various loss of strength, balance and gait disturbances arise in the central nervous system due to sensory and/or motor neuron degeneration. These disorders lead to limitations in individual activities and participation.

Fatigue is as reported one of the most common first three symptoms among patients with MS and affects up to 80% of the patients. Fatigue is defined as the lack of physical and/or mental energy. Sometimes fatigue can reduce the quality of life by leaving other disorders behind. The most important effect of fatigue is that individuals reduce their physical activity levels. This can lead to the inactivity-related secondary problems being added to the findings of the disease. So the physical capacities of individuals may gradually decrease.

In the literature, there are many studies showing that the level of physical activity of individuals with MS is lower than in healthy individuals. When the investigators analyze the studies that investigate the relation between fatigue and physical activity levels, it is seen that there is the single study about this subject in the literature.

As a result, additional studies are needed to investigate the level of physical activity and the factors affecting it in individuals with MS. Therefore, the investigators planned this study to investigate the relationship between fatigue and physical activity levels in patients with MS.

DETAILED DESCRIPTION:
According to sample size calculation 37 diagnosed Multiple Sclerosis patients and 37 healthy individuals will be included.The demographic characteristics of the participants initially will be taken and Expanded Disability Status Scale score of those of MS will be recorded. Then, fatigue severity and perception, physical activity level, balance, peripheral muscle strength, functional mobility, functional exercise capacity will be evaluated. Primary outcomes are fatigue and physical activity level; secondary outcomes are balance, peripheral muscle strength, functional mobility, functional exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Having a diagnosis of "Multiple Sclerosis" by a specialist physician
* Relapse free in the last 3 mounts
* Having an ambulatory status (Expanded Disability Status Scale score ≤ 6 )
* No diagnosis of depression

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing and perception problems that may affect the results of the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Power analysis was performed using "G * Powerversion3.1 program" in order to determine the minimum number of subjects to be taken into operation. Accordingly, the number of participants in the study group (n) = 37 (α: 0.05, for power 80%) and in the control group (n) = 37).
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Fatigue severity | Five minutes
  Fatigue Severity Scale
Fatigue | Eight minutes
  Fatigue Impact Scale
Physical activity behavior | Three days
  Evaluated using an ActiGraph (GT3X+)
Physical activity | Five minutes
  International Physical Activity Questionnaire

SECONDARY OUTCOMES:
Functional exercise capacity | Fifteen minutes
  Evaluated using 6-minute walking test
Balance | Fifteen minutes
  Evaluated using Bio Sway [(BSS) Biodex Inc.,Shirley, New York]
Functional Mobility | Two minutes
  Evaluated using Time and Go test
Muscle strength | Fifteen minutes
  Evaluated using digital hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Kader Çekim, Pt, Study Chair — Research assistant; Arzu Güçlü Gündüz, Pt, Phd, Study Director — Associate professor; Ceyla İrkeç, MD, Prof, Principal Investigator — Professor
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared

REFERENCES:
- See also: related info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Is+Physical+Behavior+Affected+in+Fatigued+Persons+With+Multiple+Sclerosis%3F
- See also: related info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Measuring+Activity+Patterns+Using+Actigraphy+in+Multiple+Sclerosis